CLINICAL TRIAL: NCT02388204
Title: Spinal Cord Stimulation for the Treatment of Motor and Nonmotor Symptoms of Parkinson's Disease
Acronym: SCSPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Erich Talamoni Fonoff, Professor of Neurosurgery, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USaoPaulo1
Record Dates: First submitted 2015-03-08; First posted 2015-03-13 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson's Disease
Keywords: Gait; Locomotion; Freezing
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parkinson's disease patients (Experimental): Group description: PD patients with locomotion problems as the primary complain with no interventions other than medication and rehabilitation therapies Intervention: Implantable spinal cord stimulation.
  Interventions: Procedure: Implantable spinal cord stimulation
- DBS Parkinson's disease patients (Experimental): Group description: PD patients with locomotion problems as the primary complain after cardinal symptoms are controlled by DBS.
  Intervention: Implantable spinal cord stimulation.
  Interventions: Procedure: Implantable spinal cord stimulation

INTERVENTIONS:
Procedure: Implantable spinal cord stimulation — Implantation of SCS electrode and pulse generator
  Other Names: Implantable SCS electrode and IPG (Medtronic)
  Arms: DBS Parkinson's disease patients
Procedure: Implantable spinal cord stimulation — Implantation of SCS electrode and pulse generator
  Other Names: Implantable SCS electrode and IPG (Medtronic)
  Arms: Parkinson's disease patients

SUMMARY:
Although DBS improves patient's quality of life advanced Parkinson's patients (PD) by addressing the cardinal symptoms and reducing levodopa motor complications, symptoms still worsen over time. Postural problems, frequent falls, freezing of gait impairment and other locomotion difficulties still remain as important causes of disability and incapacity. Novel therapeutics approaches are needed to restore quality of life (QoL).

This study aims to explore the effects of spinal cord stimulation in locomotion, falls and freezing of gait in advanced PD patients.

Twenty PD patients will undergo thoracic spinal cord stimulation at high frequencies in a prospective study for six months.

Changes in locomotion capacity and freezing of gait rating will be the primary out come. Secondary outcomes will be: QoL and common motor outcome measures in PD patients. Always comparing the status before, one, three and six months after stimulation was initiated. A double blind trial will be performed within three months of follow up (high X low frequency stimulation).

DETAILED DESCRIPTION:
Background: Currently there are no available Parkinson's disease (PD) therapy can really stop disease progression. Although Deep Brain Stimulation (DBS) improves patient's quality of life by addressing the cardinal symptoms and reducing Levodopa motor complications, non motor symptoms still increasing over time. Gait problems as falls and freezing are important cause of disability and incapacity. Novel therapeutics approaches are needed to restore quality of life. Data from animal PD model suggest that spinal cord stimulation (SCS) can enhance locomotion in mice. Although clinical results, mostly from case reports, in PD patients are still conflicting, a few patients benefited from SCS in thoracic levels.

Aim: Evaluated Spinal cord stimulation effects in locomotion, gait, freezing and falls in PD patient's.

Method: 20 PD patients will undergo thoracic spinal cord stimulation with high frequency in a prospective study for six months. Gait and freezing evaluation will consists in: timed up and go test, timed up and go test with dual task, 20 m walk test, 20 m walk test with obstacle, freezing of gait scale and falls scale. PDQ 39 and Schwab and England scales will be used to measure quality of life. Unified Parkinson's Disease Rating Scale for motor symptoms and general evaluation. All tests will be done before surgery, after one week, one, three, six months. All patients will be stimulated with the same parameters: High frequencies and 90 mcs pulse width and the sensory threshold will be measured. At the third month the parameters of SCS will be changed and comparative tested for low frequency in a double blind trail.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic PD
2. Gait and locomotion problems as the main complain/symptom
3. PD patients with or without DBS
4. Hoehn and Yahr scale equal or more than 2.0

Exclusion Criteria:

1. Dementia
2. Hoehn and Yahr scale more than 4
3. Less than 5 years of Parkinson's disease symptoms
4. General contraindications of surgery

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes in locomotion capacity | 6 months
  "Timed-up-go" test : time to complete the test : difference between scores pre-implantation and 6 months after stimulation initiation "20 meters walking test": time and steps numbers to complete the test "20 meters walking test- with obstacles": time and steps numbers to complete the test : difference between scores pre-implantation and 6 months after stimulation initiation "Dual task Timed-up-go" test : time to complete the test : difference between scores pre-implantation and 6 months after stimulation initiation "Dual task Timed-up-go" test : time to complete the test : difference between scores pre-implantation and 6 months after stimulation initiation

SECONDARY OUTCOMES:
Changes in freezing of Gait | 6 months
  FOG (freezing of gait scale): difference between scores pre-implantation and 6 months after stimulation initiation
Changes in quality of life | 6 months
  Parkinson Disease Questionnaire 39: difference between scores pre-implantation and 6 months after stimulation initiation
Motor changes | 6 months
  Unified Parkinson's Disease Rating Scale motor score: difference between scores pre-implantation and 6 months after stimulation initiation

CONTACTS AND LOCATIONS:
Overall Officials: Erich T Fonoff, MD/PhD/Prof, Principal Investigator — University of São Paulo, Department of Neurology
Locations (1):
- Division of Functional Neurosurgery, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Fuentes R, Petersson P, Nicolelis MA. Restoration of locomotive function in Parkinson's disease by spinal cord stimulation: mechanistic approach. Eur J Neurosci. 2010 Oct;32(7):1100-8. doi: 10.1111/j.1460-9568.2010.07417.x. PMID 21039949
- [Background] Fuentes R, Petersson P, Siesser WB, Caron MG, Nicolelis MA. Spinal cord stimulation restores locomotion in animal models of Parkinson's disease. Science. 2009 Mar 20;323(5921):1578-82. doi: 10.1126/science.1164901. PMID 19299613
- [Result] Agari T, Date I. Spinal cord stimulation for the treatment of abnormal posture and gait disorder in patients with Parkinson's disease. Neurol Med Chir (Tokyo). 2012;52(7):470-4. doi: 10.2176/nmc.52.470. PMID 22850494
- [Result] Fenelon G, Goujon C, Gurruchaga JM, Cesaro P, Jarraya B, Palfi S, Lefaucheur JP. Spinal cord stimulation for chronic pain improved motor function in a patient with Parkinson's disease. Parkinsonism Relat Disord. 2012 Feb;18(2):213-4. doi: 10.1016/j.parkreldis.2011.07.015. Epub 2011 Aug 23. No abstract available. PMID 21865071
- [Result] Hassan S, Amer S, Alwaki A, Elborno A. A patient with Parkinson's disease benefits from spinal cord stimulation. J Clin Neurosci. 2013 Aug;20(8):1155-6. doi: 10.1016/j.jocn.2012.08.018. Epub 2013 Feb 26. PMID 23453160
- [Result] Landi A, Trezza A, Pirillo D, Vimercati A, Antonini A, Sganzerla EP. Spinal cord stimulation for the treatment of sensory symptoms in advanced Parkinson's disease. Neuromodulation. 2013 May-Jun;16(3):276-9. doi: 10.1111/ner.12005. Epub 2012 Dec 10. No abstract available. PMID 23227965
- [Result] Thevathasan W, Mazzone P, Jha A, Djamshidian A, Dileone M, Di Lazzaro V, Brown P. Spinal cord stimulation failed to relieve akinesia or restore locomotion in Parkinson disease. Neurology. 2010 Apr 20;74(16):1325-7. doi: 10.1212/WNL.0b013e3181d9ed58. No abstract available. PMID 20404313